CLINICAL TRIAL: NCT00083265
Title: Association Between Adenosine Receptor Gene Polymorphisms and Physiological Responses to Caffeine in Subjects With Panic Disorder and Healthy Controls
Brief Title: Genetic Causes of Panic Disorder
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040183; 04-M-0183
Record Dates: First submitted 2004-05-15; First posted 2004-05-17 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02-14

CONDITIONS: Panic Disorder
Keywords: Adenosine Receptor; Panic Disorder; Polymorphism; Challenge Study; Caffeine; Healthy Volunteer; HV
MeSH Terms: conditions — Panic Disorder

SUMMARY:
This study will try to identify genes that increase the risk of developing panic disorder-an anxiety disorder characterized by recurrent unexpected panic attacks-and that contribute to the abnormalities associated with it. It will compare reactions in patients with panic disorder and in normal volunteers to caffeine, a compound that can induce anxiety, and to placebo, an inactive substance. Caffeine is believed to induce anxiety by blocking proteins called adenosine receptors on the surface of nerve cells in the brain. One study found that people with a specific adenosine receptor gene called 1976T/T had greater anxiety in response to caffeine challenge than did people with other adenosine receptor gene groups. There is also evidence that people with the 1976T/T genotype are more vulnerable to having panic disorder.

Normal volunteers and patients with panic disorder (with or without agoraphobia) who are between 18 and 60 years of age may be eligible for this study. Candidates are screened with physical and psychiatric examinations, a diagnostic interview, mood and anxiety ratings, an electrocardiogram, and blood and urine tests, including genetic studies.

Participants have two caffeine/placebo challenge sessions at least 3 days apart. Each session lasts about 4 hours. For at least 1 week before each session, subjects follow a diet excluding foods with caffeine and refrain from drinking alcoholic beverages for at least 48 hours before the procedure. The morning of the session, following an overnight fast, subjects swallow either a placebo capsule or a caffeine capsule that is equivalent to about 5 cups of coffee. During the session, subjects take a battery of neuropsychological tests to document changes in cognitive and emotional functioning, including attention, memory, and motor performance. In addition, heart rate and blood pressure are measured 15 minutes before and 30, 60, 90, 120, 150, and 180 minutes after the caffeine or placebo dose.

At the end of the study, patients with panic disorder are eligible to receive routine clinical treatment for up to 3 months and may participate in planning for long-term treatment under the care of their local health care provider.

...

DETAILED DESCRIPTION:
Caffeine, the most widely used psychoactive drug in the world, exerts its behavioral effects by antagonizing adenosine receptors (AR). Four different human AR subtypes have been found and there is evidence that the stimulatory effect of caffeine is mainly caused by an inhibition of transmission via adenosine A(2a) receptors. A significant association has been found in healthy infrequent caffeine users between caffeine-induced anxiety and two linked polymorphisms on the A(2a) receptor gene, the 1976C greater than T and 2592C greater than Tins polymorphisms. In one study looking at monozygotic and dizygotic twin pairs, there was much evidence that individual differences in caffeine use, intoxication, tolerance, and withdrawal were substantially influenced by genetic factors. Family and twin studies have shown that genetic factors may increase vulnerability to panic disorder. In one study a systematic mutation screening and association study of the A(1) and A(2a) adenosine receptor genes in panic disorder showed a significant association between the 1976T allele and 1976T/T genotype of the A(2a) receptor gene and panic disorder. As the 1976T/T genotype of the A(2a) receptor gene has been associated with both increased caffeine-induced anxiety in healthy controls, and has been associated with increased vulnerability to panic disorder, we wish to study whether the 1976T/T genotype in panic disorder patients is associated with increased caffeine-induced anxiety.

This study will study subjects with panic disorder and healthy controls. Based on previous studies the following hypotheses will be tested (2 replication and 2 new hypotheses): Replication; (1) panic disorder subjects will report higher anxiety after a caffeine challenge than the healthy control subjects. (2) healthy controls with the1976 T/T polymorphism will report increased anxiety after a caffeine challenge compared to healthy controls with the 1976 C/T and 1976 C/C genotypes, New hypotheses; (3) panic patients (two separate groups: currently ill and remitted) with the 1976 T/T polymorphism will report increased anxiety after a caffeine challenge compared to panic patients with the 1976 C/T and 1976 C/C genotypes, (4) panic patients (two separate groups: currently ill and remitted) with the 1976 T/T polymorphism will report increased anxiety after a caffeine challenge compared to healthy controls with the 1976 T/T polymorphism will report increased anxiety after a caffeine challenge compared to healthy controls with the 1976 T/T genotype.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Male or female subjects between ages 18 to 60.
  2. Panic patients with a primary diagnosis of current Panic Disorder without Agoraphobia (300.01) or Panic Disorder with Agoraphobia (300.21) according to DSM-IV criteria. Patients with co-morbid Major Depressive Disorder will be included provided there has been a period of at least 3 months where Panic Disorder, was present in the absence of Major Depressive Disorder or Patients with a past history of Panic Disorder, currently in remission. Remission is defined by as not meeting criteria for Panic Disorder for at least 3 months (no panic attacks in 3 months and less than 5 PDSS score for past month) and off treatment for at least 3 months immediately prior to study entry.
  3. Subjects must be competent to comprehend the purpose of the study and provide written informed consent.
  4. If female, subjects must be: postmenopausal, surgically incapable of childbearing, or practicing medically acceptable method(s) of contraception (eg, hormonal intrauterine device), for at least one month prior to study entry and throughout the study.
  5. Subjects must be psychotropic medication free for at lest 14 days prior to the caffeine/placebo challenge sessions; for fluoxetine at least 4 weeks.
  6. Caffeine free diet for at least 7 days prior to the caffeine/placebo challenge sessions.

EXCLUSION CRITERIA:

1. Subjects should have no general medical illness that is causing the panic disorder.
2. Serious, unstable illnesses including hepatic, renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, neurologic, immunologic, or hematologic disease.
3. Subjects with known cardiac disease.
4. Subjects with one or more past seizures without a clear and resolved etiology.
5. Patients who would be unable to comply with study procedures or assessments.
6. Patients who are currently at high risk for homicide or suicide.
7. Patients with psychotic features.
8. Patients with current DSM-IV substance abuse or dependence within the past year.
9. Patients who are on a non-psychotropic medication with psychotropic effects (e.g., beta-adrenergic blockers) unless the dosage has been stable for a minimum of one month prior to the study.
10. Subjects with a positive HIV test result.
11. Experimental treatment in the past one month.
12. For healthy volunteers, no current or past history of any psychiatric disorder.
13. Exclude subjects taking CYP1A2 inhibitors.
14. Exclude subjects with prostatitis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 117 (Actual)
Dates: Start 2004-05-13; Study Completion 2018-02-14

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Pine, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Boulenger JP, Uhde TW, Wolff EA 3rd, Post RM. Increased sensitivity to caffeine in patients with panic disorders. Preliminary evidence. Arch Gen Psychiatry. 1984 Nov;41(11):1067-71. doi: 10.1001/archpsyc.1983.01790220057009. PMID 6497568
- [Background] Chait LD. Factors influencing the subjective response to caffeine. Behav Pharmacol. 1992 Jun;3(3):219-228. PMID 11224119
- [Background] Charney DS, Heninger GR, Jatlow PI. Increased anxiogenic effects of caffeine in panic disorders. Arch Gen Psychiatry. 1985 Mar;42(3):233-43. doi: 10.1001/archpsyc.1985.01790260027003. PMID 2983630